CLINICAL TRIAL: NCT06005714
Title: Effect of Clarithromycin or Cyclosporine on Pharmacokinetics of Deuterium Hydrobromide Ramidvir Tablets in Healthy Chinese Subjects
Brief Title: Effect of Pharmacokinetics in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: JT001-018-I
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: The Effects of Clarithromycin or Cyclosporine on Pharmacokinetics of Deuterium Hydrobromide Ramidvir Tablets in Healthy Chinese Subjects
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effects of clarithromycin on pharmacokinetics of deuterium hydrobromide ramidvir tablets (Experimental)
  Interventions: Drug: Mindeudesivir hydrobromide tablets and Clarithromycin tablets; Drug: Mindeudesivir hydrobromide tablets and Cyclosporine softgels
- The effects of cyclosporine on pharmacokinetics of deuterium hydrobromide ramidvir tablets (Experimental)
  Interventions: Drug: Mindeudesivir hydrobromide tablets and Clarithromycin tablets; Drug: Mindeudesivir hydrobromide tablets and Cyclosporine softgels

INTERVENTIONS:
Drug: Mindeudesivir hydrobromide tablets and Clarithromycin tablets — Mindeudesivir hydrobromide tablets are administered once at D1 and D4, and clarithromycin tablets are administered twice from D1 to D10.
Drug: Mindeudesivir hydrobromide tablets and Cyclosporine softgels — Mindeudesivir hydrobromide tablets are administered once at D1 and D4, and cyclosporine sofgels are administered once at D4.

SUMMARY:
This study is a single-center, open label, self-controlled phase I clinical study, to evaluate the effects of clarithromycin or cyclosporine on pharmacokinetics of deuterium hydrobromide ramidvir tablets in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old ≤ age ≤ 45 years old; Gender is not limited;
2. Weight: male ≥ 50 kg, female ≥ 45 kg; Body mass index (BMI) in the range of 19-26 kg/m2 (including 19 and 26);
3. Good health status, that is, vital signs, physical examination, laboratory tests, electrocardiogram and ultrasound examination are normal or abnormal and have no clinical significance;
4. Participants who were able to take effective contraceptive measures during the study and within 3 months after the last dose of investigational product;
5. Participants who could fully understand the purpose, content and possible adverse reactions of this study, voluntarily participate in the clinical study and sign the written informed consent form, and were able to complete the entire study process and comply with the study regulations in accordance with the requirements of the study.

Exclusion Criteria:

1. Known history of allergy to the test preparation and any of its components or related preparations;
2. Subjects with allergic diseases or allergic constitutions;
3. Those who have clear diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders, etc., and require medical intervention or other diseases that are not suitable for participating in clinical trials (such as psychiatric history, etc.);
4. Those who have donated blood or lost blood ≥ 400 mL within 3 months before enrollment, or have a history of blood product use;
5. Those who have participated in clinical trials of other drugs and taken experimental drugs within 3 months before enrollment;
6. Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health supplements within 2 weeks before screening;
7. Those who have used any vaccine within 2 weeks prior to screening.
8. Those who have previously undergone surgery (such as major gastrectomy surgery) that may affect drug absorption, distribution, metabolism, or excretion, or may have surgery or hospitalization plans during the estimated test;
9. Those with a history of drug dependence or abuse within 1 year before screening, or a positive urine drug screening test;
10. Those who have used P-gp or BCRP strong inhibitors within 2 weeks before screening (see Annex 6 of Section 10.6 for details);
11. Those who have ingested grapefruit juice/grapefruit juice, foods or drinks rich in methylxanthines (such as coffee, tea, cola, chocolate, functional drinks) within 48 hours before administration, or strenuous exercise and other factors that affect drug absorption, distribution, metabolism, excretion and other factors;
12. Alcohol addict within 1 year prior to screening, drinking at least 2 times a day or more than 14 units per week, or keen on alcoholism (1 unit≈ 200 mL of beer with 5% alcohol or 25 mL of spirits with 40% alcohol or 85 mL of wine with 12% alcohol);
13. Those who smoked cigarettes within 1 year before screening, and smoked more than 10 cigarettes or the same amount of tobacco per day;
14. Those who cannot quit smoking or alcohol during the trial;
15. Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), treponemal antibody and HIV antibody positive;
16. Chest X-ray (positive and lateral view) results are abnormal and clinically significant;
17. At screening or baseline alanine aminotransferase (ALT) or glutamate aminotransferase (AST) exceeding the upper limit of normal (ULN);
18. Glomerular filtration rate (eGFR) at screening or baseline < 80 mL/min/1.73m2;
19. Abnormal ECG at screening or baseline, a single QTcF (mean of QT interval corrected by Fridericia formula) > 450 ms for men and 470 ms >for women, and/or other abnormalities of clinical significance;
20. Pregnant or lactating women or male subjects' spouses who have childcare plans within 3 months;
21. Those who have other factors that the investigator believes are not suitable for participation in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
AUC0-t of 116-N1 | At pre-defined intervals up to 14 days
  Area under the curve from time zero to the time of the t(AUC0-t ) of 116-N1
Maximum Plasma Concentration (Cmax) of 116-N1 | At pre-defined intervals up to 14 days
  Maximum Plasma Concentration (Cmax) of 116-N1

SECONDARY OUTCOMES:
Half-life(T1/2) of 116-N1 | At pre-defined intervals up to 14 days
  Half-life(T1/2) of 116-N1
Clearance(CL) of 116-N1 | At pre-defined intervals up to 14 days
  Clearance(CL) of 116-N1
Tmax of 116-N1 | At pre-defined intervals up to 14 days
  Peak time of 116-N1
Vz/F of 116-N1 | At pre-defined intervals up to 14 days
  Apparent volume of distribution of 116-N1
Incidence and severity of adverse events including serious adverse events | Up to 18 days
  Abnormal changes in clinical symptoms, vital signs, physical examination, laboratory tests, electrocardiograph and other examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Li, Principal Investigator — Zhengzhou Sixth People's Hospital
Locations (1):
- Zhengzhou Sixth People's Hospital, Zhengzhou, Henan, China